CLINICAL TRIAL: NCT05036629
Title: Development of MRI Protocols and Associated Neuro-physiological Explorations in Healthy and Pathological Subjects
Acronym: MAP-IRMaGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC20.395; 2020-A03555-34 (Other: ID RCB)
Record Dates: First submitted 2021-08-24; First posted 2021-09-05 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: MRI; Sequence Optimization; Physiological Measurement

STUDY DESIGN:
Intervention Model Description: Exploratory individual statistical analyzes on MRI data functional. No group analysis possible on these updates of MRI protocols
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI protocol (Experimental): Feasibility and use of methods developed in clinical research protocols or cognitive: the reproducibility of the parameters of acquisition, of the design of the activation paradigms development and results according to people will be an important element for the future integration of these methods in clinical or cognitive research protocols.
  Interventions: Device: MRI Protocol

INTERVENTIONS:
Device: MRI Protocol — Eye-tracker Eyelink (eye movements) BIOPAC : (electrodermal resistance) INVIVO Precess : breathing, arterial pressure, pulse,
  * NIRS Oxymon artinis medical system
  * tES (transcranial electrical stimulation, Neuroelectrics)
  Other Names: Physiological measurement during MRI protocol

SUMMARY:
IRMaGe is a Joint Service Unit (UMS) which provides users of brain exploration equipment (clinical MRI and preclinical, TMS, EEG, NIRS and metabolomics). The methods available on this equipment are intended to evolve according to the most recent discoveries and this protocol aims to frame the developments necessary around clinical MRI for IRMaGe can continue to offer tools at the cutting edge of technology.

DETAILED DESCRIPTION:
The studies will be carried out on healthy subjects and voluntary patients, who will have given their consent. Their main objective will be the development and optimization of sequence parameters or design stimulation paradigms in order to optimize the quality and relevance of the images produced taking into account the parameters anatomical, functional or metabolic while respecting the experimental constraints imposed by the protocol concerned (equipment of experimentation, additional physiological measurements, etc.). The main judgement criteria will be measurements inherent in the MRI sequence and a physiological measurement associated in the protocol concerned

ELIGIBILITY:
Inclusion Criteria:

* Participants with normal or corrected vision
* Participants affiliated to a social security scheme or beneficiaries of such a scheme
* Participants with French as their mother tongue
* Participants who have given the signed informed consent before carrying out any procedure related to the study.
* Volunteer patients will be recruited as part of their follow-up at the CHU. Their pathology will be in agreement with that of the research protocol to be optimized.

Exclusion Criteria:

Criteria relating to contraindications to the explorations provided for by the MRI protocol:

* metallic glitter in the eyes
* retinal operation
* claustrophobia
* wearer of pacemaker or cardiac defribrillator or vascular clip or prosthesis cardiac or insulin pump or implanted device to deliver medication or hearing implant or prosthesis or vascular shunt or paragraph or screws, plate metal or tattoo or piercing or implanted metal object or lead shot hunt

  * Alcohol ingestion before the examination
  * Pregnant, lactating and parturient women
  * Major protected by law
  * Participants under administrative or judicial supervision
  * Participation in another ongoing study if the study may interfere with participation in the protocol MAP-IRMaGe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2026-09-08 (Estimated); Study Completion 2026-09-08 (Estimated)

PRIMARY OUTCOMES:
Diffusion Tensor Imaging Images | 1 to 3 hours
  DTi sequences on IRM Achieva 3.0T dStream Philips
BOLD Signal | 1 to 3 Hours
  EPI sequences during cognitive protocol on IRM Achieva 3.0T dStream Philips
Anatomical Images | 1 to 3 hours
  Anatomical MR sequences on IRM Achieva 3.0T dStream Philips

SECONDARY OUTCOMES:
Eye movements | During MRI session
  Acquired by using eye-tracker (Eye-tracker Eyelink) breathing arteries pressure electrodermal conductance
Electrodermal resistance | During MRI session
  Acquired on BIOPAC device allowing physiological measurements
Blood Pressure/pulse/Breathing | During MRI session
  Acquired on INVIVO Precess
Near-infrared spectroscopy (NIRS) : Hb OHb concentration measurement | During MRI session
  Acquired with NIRS Oxymon artinis medical system
tES | During MRI session
  Transcranial Electrical stimulation, Neuroelectrics

CONTACTS AND LOCATIONS:
Locations (1):
- Unité Mixte de Service IRMaGe US 017, La Tronche, France

IPD SHARING:
Plan to Share IPD: No